CLINICAL TRIAL: NCT01444313
Title: Prospective Study of the Health Benefits of Ultra-Violet Filtering Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CR-201009
Record Dates: First submitted 2011-08-30; First posted 2011-09-30 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2014-10

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- nelfilcon A OD / narafilcon A OS (Other): Soft contact lens without UV protection worn on the right eye (OD) and soft contact lens with UV protection worn on the left eye (OS).
  Interventions: Device: narafilcon A contact lens; Device: nelfilcon A soft contact lenses
- narafilcon A OD / nelfilcon A OS (Other): Soft contact lens with UV protection worn on the right eye (OD) and soft contact lens without UV protection worn on the left eye (OS).
  Interventions: Device: narafilcon A contact lens; Device: nelfilcon A soft contact lenses

INTERVENTIONS:
Device: narafilcon A contact lens — Soft contact lenses with UV protection
Device: nelfilcon A soft contact lenses — Soft contact lenses without UV protection

SUMMARY:
The purpose of this study is to examine the short-term protective effect of Ultra-Violet filtering contact lenses on macular pigment ocular density.

ELIGIBILITY:
Inclusion Criteria:

* The subject is an adapted soft contact lens wearer
* The subject's spherical error equivalent (Best Sphere corrected for back vertex distance) must be from -0.50 diopters (D) to -6.00D or from +0.50D to +4.00D in each eye
* The subject must have a refractive astigmatism in each eye of -0.75D or less
* The subject must have a best corrected visual acuity of 6/9 or better in each eye.
* The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol
* The subject must read and sign the statement of informed consent
* The subject must be at least 18 years of age

Exclusion Criteria:

* Systemic or ocular allergies which might interfere with contact lens wear
* Systemic disease which might interfere with contact lens wear
* Ocular disease which might interfere with contact lens wear
* Grade 3 or 4 Slit Lamp Findings
* Greater than 0.1 difference in macular pigment optical density (MPOD) findings between right and left eye at baseline visit
* On changing stable medication or taking any medication known to affect tear film
* Active ocular surface pathology
* Use ocular medication
* Had had any anterior ocular surgery or other ocular surgery or injury within 8 weeks immediately prior to enrollment for this study
* Significant ocular tissue anomaly
* Presence of two or more corneal scars in either eye
* Pregnancy or lactation, or intends to become pregnant during the time period of the study
* Any medical condition that may be prejudicial to the study
* Diabetes
* Infectious diseases (e.g. Hepatitis, tuberculosis)
* Contagious immunosuppressive diseases (e.g. HIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Macular Pigment Optical Density at 9 months | baseline to 9 months
Macular Pigment Optical Density at 15 months | baseline to 15 months

SECONDARY OUTCOMES:
Macular Pigment Optical Density at 3 months | baseline to 3 months
Macular Pigment Optical Density at 6 months | baseline to 6 months
Macular Pigment Optical Density at 12 months | baseline to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Birmingham, West Midlands, United Kingdom